CLINICAL TRIAL: NCT00439075
Title: Randomised Controlled Comparison of Continuous Positive Airway Pressure (CPAP) With Standard Treatment in Out-of-hospital Patients With Acute Cardiogenic Pulmonary Edema.
Brief Title: OUT-OF-HOSPITAL CPAP STUDY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0508703
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Acute Cardiogenic Pulmonary Edema
Keywords: pulmonary disease; CPO; CPAP; oxygenation; out-of-hospital intervention
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP (Experimental): positive airway pressure
  Interventions: Procedure: CPAP
- standard medical therapy (Active Comparator): conventional oxygen therapy
  Interventions: Drug: standard treatment

INTERVENTIONS:
Procedure: CPAP
  Arms: CPAP
Drug: standard treatment
  Arms: standard medical therapy

SUMMARY:
Evaluate efficacy and safety of CPAP in a randomised standard treatment controlled study, in out-of-hospital patients with acute cardiogenic pulmonary edema.

DETAILED DESCRIPTION:
Acute cardiogenic pulmonary edema is a frequent medical emergency. Several studies have shown that continuous positive airway pressure is effective in acute cardiogenic pulmonary edema, through improvement in gas exchange, reduction in intubation rate and a trend towards reduced mortality. CPAP is usually obtained with a hermetic nasal or facemask witch has an expiratory valve to maintain a positive pressure at the end of the expiration. With this support, the patient does not receive any assistance with respiration.

The available data about CPAP concern patients hospitalised in cardiology intensive care units, in resuscitation areas or in emergency departments.

We will undertake a controlled prospective randomised trial to investigate whether the early use of CPAP would improve oxygenation and survival, as compared with standard medical therapy in patients with acute cardiogenic pulmonary edema.

This study will include 124 patients over 18 years of age, suffering of acute cardiogenic pulmonary edema, with a respiratory rate greater than 25 bpm and oxygen saturation less than 90 %. The patients will be include just after the beginning of the episode, in prehospital mobile intensive car unit (SAMU) and will be all admitted in resuscitation area in a central hospital. They will be randomly assigned to CPAP or conventional oxygen therapy. The randomisation sequence is generated by the random numbers table. Closed envelopes containing the allocated treatment will be stored in the emergency department and will be opened when the patient is included.

Oxygen saturation (by pulse-oxymetry), heart rate, respiratory rate, dyspnea, blood pressure will be measured every 15 min during the transport to the intensive care unit and every hour. The blood gazes will be measured at the arrival. The intubation rate, the duration of the hospitalisation and the mortality in the thirty days following initial treatment will be noted.

ELIGIBILITY:
Inclusion Criteria:

* patient with supposed acute cardiogenic pulmonary edema, defined as acute dyspnea associated with a past of cardiomyopathy ischemia and physical signs consistent with pulmonary edema.
* patient giving written informed consent

Exclusion Criteria:

* Glasgow score < 10
* Acute myocardial infarction ; ventricular arrhythmia ; pneumothorax ; evidence of pneumonia ; immediate need for intubation ; heart failure or respiratory stop witch requires a reanimation ; cardiogenic shock (systolic blood pressure < 90 mmhg)
* Any neurological impairment that would prevent the protocol compliance
* participation in another study throughout this one
* women pregnant or nursing
* vomiting
* patient with an history of gastric surgery (< 8days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2006-10 (Actual); Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Treatment success after the one hour study period, defined as all of respiratory rate less than 25 bpm, oxygen saturation greater than 90 %. | One hour

SECONDARY OUTCOMES:
Physiological parameters: vital signs, dyspnea , intubation rate | one hour
Safety parameters: adverse events , duration of hospitalisation , mortality 5 days and 30 days after the end of the one hour study period. | during hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: DUCASSE Jean-Louis, Principal Investigator — University Hospital, Toulouse
Locations (1):
- SAMU - University Hospital Toulouse, Toulouse, France

REFERENCES:
- [Background] Crane SD, Elliott MW, Gilligan P, Richards K, Gray AJ. Randomised controlled comparison of continuous positive airways pressure, bilevel non-invasive ventilation, and standard treatment in emergency department patients with acute cardiogenic pulmonary oedema. Emerg Med J. 2004 Mar;21(2):155-61. doi: 10.1136/emj.2003.005413. PMID 14988338
- [Background] Bellone A, Monari A, Cortellaro F, Vettorello M, Arlati S, Coen D. Myocardial infarction rate in acute pulmonary edema: noninvasive pressure support ventilation versus continuous positive airway pressure. Crit Care Med. 2004 Sep;32(9):1860-5. doi: 10.1097/01.ccm.0000139694.47326.b6. PMID 15343013
- [Background] Mehta S, Jay GD, Woolard RH, Hipona RA, Connolly EM, Cimini DM, Drinkwine JH, Hill NS. Randomized, prospective trial of bilevel versus continuous positive airway pressure in acute pulmonary edema. Crit Care Med. 1997 Apr;25(4):620-8. doi: 10.1097/00003246-199704000-00011. PMID 9142026
- [Background] L'Her E, Duquesne F, Paris A, Mouline J, Renault A, Garo B, Boles JM. [Spontaneous positive end-expiratory pressure ventilation in elderly patients with cardiogenic pulmonary edema. Assessment in an emergency admissions unit]. Presse Med. 1998 Jun 20;27(22):1089-94. French. PMID 9767807
- [Background] Evans TW. International Consensus Conferences in Intensive Care Medicine: non-invasive positive pressure ventilation in acute respiratory failure. Organised jointly by the American Thoracic Society, the European Respiratory Society, the European Society of Intensive Care Medicine, and the Societe de Reanimation de Langue Francaise, and approved by the ATS Board of Directors, December 2000. Intensive Care Med. 2001 Jan;27(1):166-78. doi: 10.1007/s001340000721. No abstract available. PMID 11280630
- [Background] Pang D, Keenan SP, Cook DJ, Sibbald WJ. The effect of positive pressure airway support on mortality and the need for intubation in cardiogenic pulmonary edema: a systematic review. Chest. 1998 Oct;114(4):1185-92. doi: 10.1378/chest.114.4.1185. PMID 9792593
- [Background] Lenique F, Habis M, Lofaso F, Dubois-Rande JL, Harf A, Brochard L. Ventilatory and hemodynamic effects of continuous positive airway pressure in left heart failure. Am J Respir Crit Care Med. 1997 Feb;155(2):500-5. doi: 10.1164/ajrccm.155.2.9032185.
- [Background] The treatment of heart failure. Task Force of the Working Group on Heart Failure of the European Society of Cardiology. Eur Heart J. 1997 May;18(5):736-53. doi: 10.1093/oxfordjournals.eurheartj.a015339. No abstract available. PMID 9152644
- [Result] Frontin P, Bounes V, Houze-Cerfon CH, Charpentier S, Houze-Cerfon V, Ducasse JL. Continuous positive airway pressure for cardiogenic pulmonary edema: a randomized study. Am J Emerg Med. 2011 Sep;29(7):775-81. doi: 10.1016/j.ajem.2010.03.007. Epub 2010 May 1. PMID 20825901